CLINICAL TRIAL: NCT05907954
Title: (Neo)Adjuvant IDE196 (Darovasertib) in Patients With Localized Ocular Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE196-009
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma; Plaque brachytherapy; Enucleation; Neoadjuvant; Adjuvant; Protein Kinase C; Ophthalmology; Ocular Oncology; Darovasertib; IDE196; Ocular melanoma; Choroid melanoma; Plaque; Brachytherapy
MeSH Terms: conditions — Uveal Melanoma; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- darovasertib (Experimental): IDE196 (darovasertib) oral open label
  Interventions: Drug: Darovasertib

INTERVENTIONS:
Drug: Darovasertib — Oral, potent, selective inhibitor of Protein Kinase C
  Other Names: IDE196; LXS196

SUMMARY:
Neoadjuvant/adjuvant IDE196 (darovasertib) in patients with primary uveal melanoma

DETAILED DESCRIPTION:
Phase 2 multi-center open-label IDE196 study in patients with primary uveal melanoma (UM) requiring either enucleation or plaque brachytherapy. Patients will be treated in neoadjuvant setting up to 12 months (or maximum benefit) followed by primary local therapy. An additional 6 months of adjuvant treatment may be given to some patients. All patients will have long term follow-up (up to 3 years) to assess visual outcome, disease recurrence, and development of metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Primary localized uveal melanoma requiring either enucleation or plaque brachytherapy
* Cohort 3 (patients with small UM tumors) - clinically diagnosed uveal (not iris) melanoma that is < 4 mm in thickness requiring treatment
* Able to dose orally
* ECOG Performance status of 0-1
* No other significant underlying ocular disease
* Adequate organ function
* Not pregnant/nursing or planning to become pregnant. Willing to use birth control

Exclusion Criteria:

* Previous treatment with a Protein Kinase C (PKC) inhibitor
* Concurrent malignant disease
* Active HIV infection or Hep B/C
* Malabsorption disorder
* Unable to discontinue prohibited medication
* Impaired cardiac function or clinically significant cardiac disease
* Any other condition which may interfere with study interpretation or results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and significant laboratory abnormalities | from first dose to 28 days after last dose of therapy, approximately 18 months
  Treatment emergent adverse events will be summarized by all AEs, all Grade 3-4-5 AEs, all treatment related AEs, all AEs leading to study drug modifications or discontinuations, all SAEs. Lab results will be summarized by change from baseline values, frequency of newly occurring on-treatment Grade 3 or 4 events; worst on-treatment value compared to baseline.
Cohort 1 (enucleation): Number of patients converted from requiring enucleation to radiation | from first dose of neoadjuvant to end of neoadjuvant therapy, approximately 12 months
  Rate of eye salvage as determined by the ocular oncologist based on tumor response to neoadjuvant therapy
Cohort 2 (plaque brachytherapy): Estimated change in modeled radiation dose | from first dose of neoadjuvant to end of neoadjuvant therapy, approximately 12 months
  Change in modeled radiation dose at critical eye structures before and after neoadjuvant therapy
Cohort 3 (patients with small UM tumors): Number of patients with clinical benefit per protocol-defined UM response criteria | from first dose of neoadjuvant to end of neoadjuvant therapy, approximately 12 months
  Proportion of patients with clinical benefit rate (CBR) defined as complete response (CR) + partial response (PR) + stable disease (SD) for ≥ 12 weeks per UM response criteria

SECONDARY OUTCOMES:
Evaluate tumor response to neoadjuvant IDE196 | from first dose of neoadjuvant to end of neoadjuvant therapy, approximately 12 months
  Measurement of tumor diameter and thickness before and after neoadjuvant therapy with IDE196, specifically as measured by ocular ultrasound, evaluating largest basal diameter and apical thickness of the uveal melanoma (measured in millimeters)
Assessment of visual acuity loss | from time of primary local therapy to one year after surgery, approximately 12 months
  Best corrected visual acuity loss over time
Rate of local disease recurrence | from date of primary local therapy to end of follow-up, approximately 36 months
  Evaluate uveal melanoma progression or recurrence
Cohort 3 (patients with small UM tumors): Effect of neoadjuvant IDE196 therapy on the natural history of small UM tumors | from first dose of neoadjuvant to primary local therapy, approximately 12 months
  Time from first dose of neoadjuvant to primary local therapy
Cohort 3 (patients with small UM tumors): Efficacy of neoadjuvant IDE196 therapy on small UM tumors | from first dose of neoadjuvant to end of neoadjuvant therapy, approximately 12 months
  Tumor response (complete response and partial response) as measured by protocol-defined UM response criteria

OTHER OUTCOMES:
Rate of metastatic disease | from date of primary local therapy to end of follow-up, approximately 36 months
  Evaluate occurrence of metastatic uveal melanoma
Overall survival | from date of first dose to end of follow-up, approximately 54 months
  Evaluate patient survival status

CONTACTS AND LOCATIONS:
Overall Officials: Jasgit Sachdev, MD, Study Director — IDEAYA Biosciences
Locations (24):
- United States (13):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - University of Miami, Miami, Florida
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell, Manhasset, New York
  - Duke University Health System, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - St. Vincent's Health Sydney, Sydney, New South Wales
  - Alfred Health, Melbourne, Victoria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Institute Curie, Paris, France
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Instituto Nazionale Tumori IRCCS - Fondazione Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Leiden University Medical Center, Leiden, Netherlands
- United Kingdom (2):
  - University College London Hospital - NHS Foundation Trust, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: No